CLINICAL TRIAL: NCT01464463
Title: The Impact of Psychological Interventions (With and Without Exercise) on Psychometric and Immunological Measures in Patients With Major Depression
Brief Title: The Impact of Psychological Interventions on Psychometric and Immunological Measures in Patients With Major Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Winfried Rief, Prof.Dr. / Principal investigator / Head of the department of clinical psychology and psychotherapy, Philipps University of Marburg, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFG RI 574/23-1
Record Dates: First submitted 2011-10-19; First posted 2011-11-03 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Depression
Keywords: Depression; Exercise; Psychoneuroimmunology; Cognitive Behavioral Therapy; CBASP
MeSH Terms: conditions — Depression; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CBT-active (Experimental): Patients with Major Depression (N = 50) get a common CBT treatment in combination with physical exercise.
  Interventions: Behavioral: CBT - active
- CBT-euthymic (Active Comparator): Patients with Major Depression (N = 50) get the same common CBT treatment as the CBT-active-group, but instead of physical exercise they receive an enjoyment training, which is based on exercises from the "Kleine Schule des Genießens" (Koppenhöfer, 2004)
  Interventions: Behavioral: CBT - euthymic
- CBASP (Active Comparator): Patients with Major Depression (N=50) get a cognitive therapy according to the Cognitive Behavioral Analysis System of Psychotherapy (CBASP).
  Interventions: Behavioral: CBASP
- Waiting List (No Intervention): Patients randomized to the waiting list receive psychological treatment after waiting for 4 month.

INTERVENTIONS:
Behavioral: CBT - active — Patients get CBT treatment combined with moderate physical exercise (4x40min/week for 4 weeks, week 5, 6, 7 and 8).
  Arms: CBT-active
Behavioral: CBT - euthymic — Patients get the same common CBT treatment as group I, but instead of physical exercise they receive an enjoyment training Patients get CBT treatment combined with euthymic exercise (4x40min/week for 4 weeks, week 5, 6, 7 and 8).
  Arms: CBT-euthymic
Behavioral: CBASP — Cognitive Behavioral Analysis System of Psychotherapy integrates behavioral, cognitive, psychodynamic and interpersonal strategies.
  Foci of the CBASP-therapy are situation analysis and subsequent behavioral trainings as well as interpersonal strategies to create a therapeutic relationship.
  Arms: CBASP

SUMMARY:
The objective of this study is to compare the impact of i) Cognitive Behavioral Therapy (CBT) combined with exercise, ii)CBT combined with euthymic therapy, and iii) 'Cognitive Behavioral Analysis System of Psychotherapy' (CBASP) on psychometric and immunological measures in patients with major depression.

DETAILED DESCRIPTION:
The interest of the investigation is to compare the impact of CBT combined with exercise, CBT combined with euthymic therapy and CBASP on depression and further psychopathological variables (assessed at 5 points).

Previous findings indicate increased concentration of pro-inflammatory cytokines in depression. A bidirectional relationship between depression and immunological alterations has been suggested: On the one hand pro-inflammatory cytokines may contribute to depression, on the other hand depression-linked changes (e.g. a reduction of activity, increased stress-sensitivity) may lead to increased secretion of pro-inflammatory cytokines. Therefore, this study is also supposed to investigate the influence of above mentioned interventions on pro-inflammatory cytokines. Using a waiting group, potential changes in psychometric and biological parameters without any intervention are controlled. Assessments take place at baseline, after 4 weeks of treatment, after 8 weeks of treatment, after 16 weeks of treatment and 6 months follow up.

200 patients with Major Depression (DSM IV, BDI II at baseline ≥18) will be included. Patients will be randomized and assigned to one of the 4 groups.

ELIGIBILITY:
Inclusion Criteria:

* patients with Major Depression (DSM IV), BDI >=18
* age:18-65 years
* patients with and without antidepressive medication
* comorbidity with other psychiatric disorders is permitted, as far as depressive symptoms are dominating

Exclusion Criteria:

* current psychotherapy
* psychotic disorder
* serious drug-addiction
* drugs which seriously affect immune status (except contraceptives) or central nervous system functions (except antidepressants)
* infections during the last 2 weeks
* injuries during the last 2 weeks
* neurological disorders
* diseases which affect immune status or central nervous system functions (e.g. rheumatoid arthritis, CVD,etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-08; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Changes in severity of depressive symptoms from baseline (beginning of therapy) to 4 weeks after baseline, to 8 weeks after baseline, to 16 weeks after baseline (end of therapy) to 6-month-follow up | From baseline (beginning of therapy) to 4 weeks after baseline, to 8 weeks after baseline, to 16 weeks after baseline (end of therapy) to 6-month-follow up
  Becks Depression Inventory II (BDI-II; german adaptation by Hautzinger, Kühner & Keller, 2006)

SECONDARY OUTCOMES:
Changes in immunological measures from baseline (beginning of therapy) to 4 weeks after baseline, to 8 weeks after baseline, to 16 weeks after baseline (end of therapy) to 6-month-follow up | From baseline (beginning of therapy) to 4 weeks after baseline, to 8 weeks after baseline, to 16 weeks after baseline (end of therapy) to 6-month-follow up
  C-reactive protein, inflammatory markers(Il-6, TNF-alpha, INF-gamma, IL-1ra, sTNF-RI, sTNF-RII) and anti-inflammatory cytokines (Il-10)
Changes in psychopathological variables from baseline (beginning of therapy) to 4 weeks after baseline, to 8 weeks after baseline, to 16 weeks after baseline (end of therapy) to 6-month-follow up | From baseline (beginning of therapy) to 4 weeks after baseline, to 8 weeks after baseline, to 16 weeks after baseline (end of therapy) to 6-month-follow up
  Symptom-Checklist by Derogatis (SCL-90-R; german adaption by Franke, 1995)
Changes in perceived stress from baseline (beginning of therapy) to 4 weeks after baseline, to 8 weeks after baseline, to 16 weeks after baseline (end of therapy) to 6-month-follow up | From baseline (beginning of therapy) to 4 weeks after baseline, to 8 weeks after baseline, to 16 weeks after baseline (end of therapy) to 6-month-follow up
  Trier inventary for chronic stress (TICS-K; Trierer Inventar zu chronischen Stress; Schulz et al., 2004)
Changes in self-rated physical activity from baseline (beginning of therapy) to 4 weeks after baseline, to 8 weeks after baseline, to 16 weeks after baseline (end of therapy) to 6-month-follow up | From baseline (beginning of therapy) to 4 weeks after baseline, to 8 weeks after baseline, to 16 weeks after baseline (end of therapy) to 6-month-follow up
  Internationational Physical Activity Questionaire (IPAQ, Granger et al., 2000)
Changes from baseline to 16 weeks after baseline (end of therapy) | From baseline to 16 weeks after baseline (end of therapy)
  Verbal test for learning- and memory abilities (Verbaler Lern- und Merkfähigkeitstest-VLMT; Helmstaedter, Lendt, Lux, 2001)

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Prof., Study Director — Philipps University Marburg
Locations (1):
- Department of Clinical Psychology and Psychotherapy, Philipps University Marburg, Marburg, Germany